CLINICAL TRIAL: NCT04119388
Title: Evaluation of the Benefits of Adaptive Physical Activity in Children and Adolescents With Osteogenesis Imperfecta
Acronym: MOVE-OI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL18_0747; ID-RCB (Other: 2018-A03041-54)
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: osteogenesis imperfecta; Adapted sport; Quality of life
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adapted sports practice (Experimental): patients with osteogenesis imperfect will practice adapted sport twice a week during 12 months in order to improve their aerobic capacity, cardiovascular and bone benefits, and gain of quality of life.
  Interventions: Other: Adapted sports practices

INTERVENTIONS:
Other: Adapted sports practices — Adapted sports practices for 30 minutes twice a week

SUMMARY:
Osteogenesis imperfecta (OI) is a rare genetic disorder of increased bone fragility and low bone mass. It is conceivable that children and adolescents with OI are less active than healthy peers because of frequent fractures, immobilization,functionals limitations and no adapted physicals activity(APA). The hypothesis is that an Adapted physique activity could improve access of activity for patients with Osteogenesis Imperfecta (OI).

The aim of the study is to evaluate benefice of APA,improve aerobic capacity, cardiovascular and bone benefits, and gain of quality of life.

Children with OI between 6 and 18 years old will have a program of supervised "adapted training program" during one year. The program is adapted at each individual and without risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Child with osteogenesis imperfecta
* Child followed in the Reference centre for constitutional bone diseases in the Hôpital Femme Mère Enfant
* Parent (s) / legal guardian who has been informed of the study and has accepted participation in the study by signing the consent.
* Patient benefiting from a social security scheme

Exclusion Criteria:

* Medical and surgical contraindications to adapted physical activity.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | Month 0
  Distance traveled (in meters) in 6 minutes
6 minutes walk test | Month 6
  Distance traveled (in meters) in 6 minutes
6 minutes walk test | Month 12
  Distance traveled (in meters) in 6 minutes

SECONDARY OUTCOMES:
Weight | Month 0
  weight in kilograms will be measured with a scale
Weight | Month 6
  weight in kilograms will be measured with a scale
Weight | Month 12
  weight in kilograms will be measured with a scale
Height | Month 0
  Size in meter measured with a meter
Height | Month 6
  Size in meter measured with a meter
Height | Month 12
  Size in meter measured with a meter
body mass index | Month 0
  calculated with weight and height
body mass index | Month 6
  calculated with weight and height
body mass index | Month 12
  calculated with weight and height
blood pressure | Month 0
  measurement of blood pressure (cm Hg)
blood pressure | Month 6
  measurement of blood pressure (cm Hg)
blood pressure | Month 12
  measurement of blood pressure (cm Hg)
phosphocalcic biologic parameters | Month 0 and Month 12
  Ionosodium (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  potassium (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  calcium (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  chlore (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  bicarbonates (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  glucose (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  urea (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  creatinemia (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  phosphorus (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  proteinemia (g/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  Vitamin D (nmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  1-25 OH vitamin D (pmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  PTH (ng/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  alkaline bone phosphatases (U/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  CTX (pg/ml)crosslaps
phosphocalcic biologic parameters | Month 0 and Month 12
  osteocalcin (µg/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  ferritin (µg/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  blood count formula : leucocytes (giga/L), erythrocytes (tera/L), hemoglobin (g/L), hematocrit (%), platelets (giga/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  calciuria (mmol/L)
phosphocalcic biologic parameters | Month 0 and Month 12
  Ionosodium (mmol/L) potassium (mmol/L), calcium (mmol/L), chlore (mmol/L), bicarbonates (mmol/L), glucose (mmol/L), urea (mmol/L), creatinemia (mmol/L), phosphorus (mmol/L), proteinemia (g/L), Vitamin D (nmol/L), 1-25 OH vitamin D (pmol/L), PTH (ng/L), alkaline bone phosphatases (U/L), CTX (pg/ml)crosslaps, osteocalcin (µg/L), NFS, ferritin (µg/L), blood count formula : leucocytes (giga/L), erythrocytes (tera/L), hemoglobin (g/L), hematocrit (%), platelets (giga/L), calciuria (mmol/L), urinary creatinin (mmol/L).
ration lean mass / fat mass | Month 0
  Dual-energy X-ray absorptiometry (DXA)
ration lean mass / fat mass | Month 12
  Dual-energy X-ray absorptiometry (DXA)
Respiratory Functional Exploration | Month 0
Respiratory Functional Exploration | Month 12
Thickness intima / media | Month 0
  echography
Parameters of the connected watch : number of steps | Month 0 and Month 6 and Month 12
  data recovery of the connected watch
Parameters of the connected watch : distance traveled | Month 0 and Month 6 and Month 12
  data recovery of the connected watch
Parameters of the connected watch : calories consumption | Month 0 and Month 6 and Month 12
  data recovery of the connected watch
Ratio thickness intima / media | Month 12
  echography
Bone mineral density | Month 0
  Dual-energy X-ray absorptiometry (DXA)
Bone mineral density | Month 12
  Dual-energy X-ray absorptiometry (DXA)
Number of new fractures | Month 1
Number of new fractures | Month 3
Number of new fractures | Month 6
Number of new fractures | Month 9
Number of new fractures | Month 12
Quality of life questionnaire : PedsQL | Month 0
  Measurement Model for the Pedratric Quality of Life Inventory
  The 4 Multidimensional Scales and 3 Summary Scores are
  Scales Physical Functioning (8 items) Emotional Functioning (5 items) Social Functioning (5 items) School Functioning (5 items)
  Summary Scores Total Scale Score (23 items) Physical Health Summary Score (8 items) Psychosocial Health Summary Score (15 items)
Quality of life questionnaire : PedsQL | Month 6
  Measurement Model for the Pedratric Quality of Life Inventory
  The 4 Multidimensional Scales and 3 Summary Scores are
  Scales Physical Functioning (8 items) Emotional Functioning (5 items) Social Functioning (5 items) School Functioning (5 items)
  Summary Scores Total Scale Score (23 items) Physical Health Summary Score (8 items) Psychosocial Health Summary Score (15 items)
Quality of life questionnaire : PedsQL | Month 12
  Measurement Model for the Pedratric Quality of Life Inventory
  The 4 Multidimensional Scales and 3 Summary Scores are
  Scales Physical Functioning (8 items) Emotional Functioning (5 items) Social Functioning (5 items) School Functioning (5 items)
  Summary Scores Total Scale Score (23 items) Physical Health Summary Score (8 items) Psychosocial Health Summary Score (15 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence des Maladies Rénales Rares - Hospices Civils de Lyon - Service de Néphrologie et Rhumatologie Pédiatriques - Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Arab H, Flammier S, Espitalier M, Bacchetta J, Fouillet-Desjonqueres M. Evaluation of the benefits of adapted physical activity in children and adolescents with osteogenesis imperfecta: the MOVE-OI trial. Orphanet J Rare Dis. 2025 Apr 12;20(1):175. doi: 10.1186/s13023-025-03678-4. PMID 40221747